CLINICAL TRIAL: NCT01694134
Title: Assessment of the Efficacy of an Intradiscal Injection of Corticoids in Modic I Discopathies.
Acronym: MODISC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8833
Record Dates: First submitted 2012-09-22; First posted 2012-09-26 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Low Back Pain; Lumbago; Modic I Discopathy
Keywords: Discopathy; Modic I; Corticoids; Local Anaesthetic; Intradiscal injection
MeSH Terms: conditions — Low Back Pain | interventions — Methylprednisolone; Lidocaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Corticoids (Active Comparator): A group of patients will receive an intradiscal injection of Hydrocortancyl.
  Interventions: Drug: Hydrocortancyl.
- Local anaesthetic (Sham Comparator): A group of patients will receive an intradiscal injection of Lidocaine.
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Hydrocortancyl. — Patients will receive an intradiscal injection of hydrocortancyl.
  Arms: Corticoids
Drug: Lidocaine
  Arms: Local anaesthetic

SUMMARY:
The treatment of chronic low back pain is a major objective of public healthcare, because it causes an important number of sick leaves. A correlation between clinical observations and an inflammatory discopathy has been underlined, but there is currently any reference treatment. In this study, the main objective is to assess the efficacy of an intradiscal injection of corticoids versus local anaesthetic on the treatment of pain of patients with low back pain associated to a Modic I discopathy.

DETAILED DESCRIPTION:
This is a randomized, controlled, single-blind with two arms (anaesthetic versus corticoids) trial.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years
* Signed Informed consent
* Low back pain for more than 6 months associated with Modic I discopathy (diagnosed by MRI)

Exclusion Criteria:

* Past history of lumbar surgery
* Patient under anticoagulant or antisludge treatment, or with coagulation troubles
* Patient with unbalanced diabetes mellitus (blood glucose > 1.30 g/l)
* Patient with unstabilized high blood pressure (> 160/95 mmHg)
* Patient with evolving infection
* Patient with iodine allergy or one of the Hydrocortancyl® or Lidocaine components
* Porphyria, hypersensitivity to local anaesthetic
* Patient with sphincter troubles showing a cauda equine syndrome
* Untreated psychotic state
* Pregnant women or of childbearing age without effective contraception means
* Impossible 6 months follow-up
* Participation to another trial
* Vulnerable persons protected by the law
* Persons under guardianship
* Persons unable to express their consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-07-12 (Actual); Primary Completion 2017-03-20 (Actual); Study Completion 2017-03-20 (Actual)

PRIMARY OUTCOMES:
Pain assessment: VAS | 1 month
  The pain will be assessed by the visual analog scale (VAS).

SECONDARY OUTCOMES:
Pain assessment: VAS | 1 week, 2 weeks, 3 weeks, 3 months, 6 months
  The pain will be assessed by the visual analog scale (VAS).
Quality of life assessment: SF-36 | 1 month, 3 months, 6 months
  Quality of life will be assessed by the self-questionnaire SF-36.
Consumption of analgesics and NSAIDs assessment | 1 month, 3 months,6 months
Specific low back pain parameters assessment | 1 month, 3 months,6 months
  Low back pain parameters will be assessed by the Dallas scale.The Dallas Pain Questionnaire (DPQ) assesses the impact of low back pain (LBP) on four components (0-100) of daily life .
Specific low back pain parameters assessment | 1 month, 3 months,6 months
  Low back pain parameters will be assessed by the Oswestry scale. The self-completed questionnaire contains ten topics concerning intensity of pain, lifting, ability to care for oneself, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel. Each topic category is followed by 6 statements describing different potential scenarios in the patient's life relating to the topic. The patient then checks the statement which most closely resembles their situation. Each question is scored on a scale of 0-5 with the first statement being zero and indicating the least amount of disability and the last statement is scored 5 indicating most severe disability. The scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability possible.
Employment status | 1 month, 3 months,6 months
  Employment or non-employment status will be noted

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital University of Montpellier, Montpellier, France